CLINICAL TRIAL: NCT02666053
Title: A Study to Assess the Effect of a High-fat Meal and Increased Gastric pH on the Bioavailability of an Extended-release Formulation of BMS-663068 in Healthy Subjects
Brief Title: A Study to Assess the Effect of High Fat Meal and Increased Gastric pH on the Bioavailability of an Extended Release Formulation of BMS-663068 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Other
Other Study IDs: 206295; AI438-071 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2016-01-07; First posted 2016-01-28 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): Single BMS-663068 tablet under fasted conditions
  Interventions: Drug: BMS-663068
- Treatment B (Experimental): Single BMS-663068 tablet with a high fat meal
  Interventions: Drug: BMS-663068
- Treatment C (Experimental): Single BMS-663068 tablet after a single famotidine tablet under fasted conditions
  Interventions: Drug: BMS-663068

INTERVENTIONS:
Drug: BMS-663068 — BMS-663068

SUMMARY:
The purpose of this study is to estimate the effect of high fat meal and increased gastric pH on BMS-663068 bioavailability

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Target population: Healthy males and females.
3. Males and females
4. Women of child bearing potential (WOCBP) with negative serum or urine pregnancy test
5. Women must not be breastfeeding
6. Men and WOCBP must agree to follow instructions for contraception

Exclusion Criteria:

1. History of any chronic or acute illness or gastrointestinal disease
2. Any major surgery within 4 weeks of study drug administration
3. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population.
4. History of allergy to HIV attachment inhibitors, famotidine or high fat meal
5. History of smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2016-02-22 (Actual); Study Completion 2016-02-22 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Days 1-12
Area under the plasma concentration-time curve from time zero extrapolated to infinity, AUC (INF) | Days 1-12

SECONDARY OUTCOMES:
Safety endpoints include incidence of nonserious AEs, serious AEs, AEs leading to discontinuation | Days 1-12; for SAEs up to 30 days post discontinuation of dosing
  Adverse events (both serious and nonserious) will be listed and tabulated by system organ class, preferred term, and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States